CLINICAL TRIAL: NCT04221438
Title: A Phase II Neoadjuvant Study of Encorafenib With Binimetinib in Patients With Resectable Locoregional Metastases From Cutaneous or Unknown Primary Melanoma (Stages III N1B/C/D)
Brief Title: Testing Treatment With Encorafenib and Binimetinib Before Surgery for Melanoma With Lymph Node Involvement
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA6183; NCI-2019-07407 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA6183 (Other: ECOG-ACRIN Cancer Research Group); EA6183 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Melanoma of Unknown Primary; Metastatic Malignant Neoplasm in Lymph Node; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Recurrent Cutaneous Melanoma
MeSH Terms: conditions — Lymphatic Metastasis; Melanoma | interventions — binimetinib; encorafenib; alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant encorafenib + binimetinib, surgery, adjuvant encorafenib + binimetinib (Experimental): NEOADJUVANT TREATMENT: Patients receive 18F-FLT IV and undergo a PET/CT scan approximately 60 minutes later. Within 2 weeks, patients receive encorafenib PO QD and binimetinib PO BID on days 1-28. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive 18F-FLT IV and undergo a second PET/CT scan approximately 60 minutes later.
  SURGICAL RESECTION: Within 2 weeks of completing therapy with encorafenib and binimetinib, patients undergo surgery.
  ADJUVANT TREATMENT: Within 2-7 days after surgery, patients resume treatment with encorafenib PO QD and binimetinib PO BID on days 1-28. Treatment repeats every 28 days for up to 11 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Binimetinib; Procedure: Conventional Surgery; Drug: Encorafenib; Other: Fluorothymidine F-18

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: NSC 788187; ARRY-438162; MEK162; Mektovi
Procedure: Conventional Surgery — Undergo surgery
Drug: Encorafenib — Given PO
  Other Names: ONO-7702; LGX818
Other: Fluorothymidine F-18 — Given IV
  Other Names: 18F-FLT; 3'-deoxy-3'- 18F fluorothymidine; FLT

SUMMARY:
This phase II trial studies how well encorafenib and binimetinib work before surgery in treating patients with BRAF V600-mutated stage IIIB-D melanoma that has spread to the lymph nodes. Encorafenib and binimetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This trial also studies how well 18F-FLT positron emission tomography (PET)/computed tomography (CT) works in predicting the response of melanoma to encorafenib and binimetinib. 18F-FLT is an imaging agent, sometimes called a tracer. PET and CT are types of imaging scans. Using 18F-FLT PET/CT together with encorafenib and binimetinib may provide more information on melanoma over time.

DETAILED DESCRIPTION:
PRIMARY CLINICAL OBJECTIVE:

I. To evaluate the pathologic complete response (pCR) rate of neoadjuvant treatment with encorafenib and binimetinib.

SECONDARY CLINICAL OBJECTIVES:

I. To determine response rate (RR) (Response Evaluation Criteria in Solid Tumors [RECIST]), disease-free survival (DFS) and overall survival (OS).

II. To describe correlation of pCR with RR, DFS and OS. III. To assess safety and toxicity.

CORRELATIVE SCIENCE OBJECTIVES:

I. To evaluate CD8 positive (+) T cell infiltration and Ki-67 status in tumor or tumor bed pre, during, and post neoadjuvant treatment and the change in CD8+ tumor infiltrating lymphocyte (TIL) with neoadjuvant treatment and correlate with clinical response.

II. To compare local review for pathologic response with central pathology review.

III. To assess the correlation between change in fluorothymidine F-18 (18F-FLT) PET/CT uptake and change in Ki-67.

IMAGING OBJECTIVES:

I. To compare the change in 18F-FLT PET/CT uptake (from baseline to post-neoadjuvant therapy) among patients with and without pathologic complete response.

II. To compare post-neoadjuvant 18F-FLT PET/CT uptake among patients with and without pathologic complete response.

III. To estimate an optimal threshold for prediction of pathologic complete response using i) change in 18F-FLT PET/CT uptake, and ii) post-neoadjuvant 18F-FLT PET/CT uptake.

IV. To assess the correlation between change in 18F-FLT PET/CT uptake and change in Ki-67.

OUTLINE:

NEOADJUVANT TREATMENT: Patients receive 18F-FLT intravenously (IV) and undergo a PET/CT scan approximately 60 minutes later. Within 2 weeks, patients receive encorafenib orally (PO) once daily (QD) and binimetinib PO twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive 18F-FLT IV and undergo a second PET/CT scan approximately 60 minutes later.

SURGICAL RESECTION: Within 2 weeks of completing therapy with encorafenib and binimetinib, patients undergo surgery.

ADJUVANT TREATMENT: Within 2-7 days after surgery, patients resume treatment with encorafenib PO QD and binimetinib PO BID on days 1-28. Treatment repeats every 28 days for up to 11 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically proven melanoma that is clinically evident (macroscopic lymphadenectomy [LAD]) stage III B/C/D, (American Joint Committee on Cancer [AJCC] 8th edition) of cutaneous origin or unknown primary. Patients must have at least one clinically evident lymph node metastasis (N1c patients are not eligible).

  * This may be an initial presentation with primary tumor and nodal metastases or locoregional nodal relapse with history of resected primary melanoma
  * Stage IIIB

    * T0-3a N1b M0
    * T1a-3a N2b M0
  * Stage IIIC

    * T0 or T3b-4b N2b M0
    * T3b-4b N1b M0
    * Any T N2c M0 (at least 1 clinically evident node)
    * T0-4a N3b M0
  * Stage IIID

    * T4b N3b/c M0 (if 3c: at least 1 clinically evident node)
* Patient must have measurable disease on baseline imaging scans, obtained within 4 weeks prior to registration as defined by RECIST and by the following criteria

  * The melanoma target tumor must be completely resectable as determined by a surgical oncologist or experienced melanoma surgeon

    * Extensive satellitosis or in transit metastases are not considered completely resectable
* Patient must have BRAF V600 mutation positive based on report from Clinical Laboratory Improvement Act (CLIA) certified laboratory
* Patient must be medically fit to undergo surgery
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (obtained < 14 days prior to registration)
* Hemoglobin >= 8 g/dL without transfusion (obtained < 14 days prior to registration)
* Platelets >= 100 x 10^9/L without transfusion (obtained < 14 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.0 x upper limit of normal (ULN) (obtained < 14 days prior to registration)
* Total bilirubin =< 1.5 x ULN and < 2 mg/dL; OR total bilirubin > 1.5 x ULN with indirect bilirubin < 1.5 x ULN (obtained < 14 days prior to registration)
* Serum creatinine =< 1.5 x ULN, or calculated creatinine clearance > 50 mL/min by Cockcroft-Gault formula (obtained < 14 days prior to registration)
* Prothrombin time (PT), international normalized ratio (INR), and partial thromboplastin time (PTT) =< 1.5 x ULN (obtained < 14 days prior to registration)
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patient must be able to take oral medications
* Patient must be able to lie still during the 18F-FLT PET/CT scan for the duration of the imaging study (up to 1.5 hours), have no previous indication of allergic reaction to the radiotracer, and meet the size limits of the qualified PET/CT scanner
* Patient must be participating in this study at an institution which has completed the ECOG-American College of Radiology Imaging Network (ACRIN) defined PET/CT scanner qualification procedures and received ECOG-ACRIN PET scanner approval
* Patients known to be human immunodeficiency virus (HIV) positive are eligible if they have undetectable HIV viral load and stable and adequate CD4 counts (>= 500 mm^3) on screening labs provided they meet all other protocol criteria for participation and that there is no high risk drug interactions
* Women of childbearing potential and sexually active males must use accepted and effective method(s) of contraception or to abstain from sexual intercourse for the duration of their participation in the study and for at least 30 days after the last dose of protocol treatment for female patients, and for at least 90 days after the last dose of protocol treatment for male patients. In addition, female patients must not donate ova from the time of registration until 30 days after the last dose of study treatment. Male patients must not donate sperm from the time of registration until 90 days after the last dose of protocol treatment
* Patient may be on anticoagulation at prophylactic or therapeutic levels. Patients must not be using anticoagulants at therapeutic levels that may interfere with encorafenib and binimetinib

Exclusion Criteria:

* Stage IV melanoma
* Patient must not have any prior treatment with BRAF inhibitor (BRAFi) or MEK inhibitor (MEKi)
* Patient must not have any evidence of distant metastases
* Patient must not have any prior adjuvant therapy at this disease presentation; prior immune therapy (such as adjuvant interferon or checkpoint inhibitors) is permitted if >= 6 months from last treatment
* Patient must not have any prior radiation to the site of evaluable disease
* Patient must not have active infection requiring treatment with parenteral antibiotics
* Patient must not have active hepatitis B, and/or active hepatitis C infection given concerns for drug interactions or increased toxicities. Testing is not required
* Patient must not have other significant medical, surgical, or psychiatric conditions that in the opinion of the investigator may interfere with compliance, make the administration of study medications hazardous
* Patient must not have had previous or concurrent other malignancy with the following exceptions:

  * Adequately treated basal cell or squamous cell carcinoma of the skin, in situ carcinoma of the cervix
  * Other solid tumor: if treated and without evidence of recurrence for at least 2 years prior to study entry
* Women must not be pregnant or breast-feeding due to potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the systemic antineoplastic medications, as well as surgery and radiation being used. Patients must also not expect to conceive or father children from the time of registration, while on study, treatment, and until at least 30 days after the last dose of study treatment (for female patients) and 90 days after the last dose of study treatment (for male patients). All females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient must not have known hypersensitivity or contraindication to any component of binimetinib or encorafenib or their excipients
* Patient must not have impaired cardiovascular function or clinically significant cardiovascular disease including, but not limited to, any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) < 6 months prior to registration
  * Congestive heart failure requiring treatment (New York Heart Association grade >= 2)
  * Left ventricular ejection fraction (LVEF) < 50% as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO)
  * Uncontrolled hypertension defined as persistent systolic blood pressure >= 150 mmHg or diastolic blood pressure >= 100 mmHg despite current therapy
  * History or presence of clinically significant cardiac arrhythmias (including resting bradycardia, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia)
  * Baseline corrected QT (QTc) interval >= 480 ms
* Patient must not have impairment of gastrointestinal function or disease which may significantly alter the absorption of study drug (e.g., active ulcerative disease, uncontrolled vomiting or diarrhea, malabsorption syndrome, small bowel resection with decreased intestinal absorption), or recent (=< 3 months) history of a partial or complete bowel obstruction, or other conditions that will interfere significantly with the absorption of oral drugs
* Patient must not have any known history of acute or chronic pancreatitis
* Patient must not have any concurrent neuromuscular disorder that is associated with elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy
* Patient must not have any known history or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity, factor V Leiden or activated protein C resistance); history of retinal degenerative disease
* Patient must not use any medication (including herbal medications, supplements, or foods), or use of a prohibited medication =< 1 week prior to registration
* Patient must not have a history of thromboembolic or cerebrovascular events =< 12 weeks prior to registration. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e. massive or sub-massive) deep vein thrombosis or pulmonary emboli

  * NOTE: Patients with thromboembolic events related to indwelling catheters or other procedures may be registered
  * NOTE: Patients with either deep vein thrombosis or pulmonary emboli that does not result in hemodynamic instability are allowed to register as long as they are on a stable dose of anticoagulants for at least 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Fecher, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (10):
- United States (10):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on February 18, 2020 and the first patient was enrolled in September, 2021. The study was closed on September 23, 2022 due to slow accrual.
Groups:
- Experimental: Neoadjuvant Encorafenib + Binimetinib, Surgery, Adjuvant Encorafenib + Binimetinib: NEOADJUVANT TREATMENT: Patients receive 18F-FLT IV and undergo a PET/CT scan approximately 60 minutes later. Within 2 weeks, patients receive encorafenib PO QD and binimetinib PO BID on days 1-28. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive 18F-FLT IV and undergo a second PET/CT scan approximately 60 minutes later.
  SURGICAL RESECTION: Within 2 weeks of completing therapy with encorafenib and binimetinib, patients undergo surgery.
  ADJUVANT TREATMENT: Within 2-7 days after surgery, patients resume treatment with encorafenib PO QD and binimetinib PO BID on days 1-28. Treatment repeats every 28 days for up to 11 cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Experimental: Neoadjuvant Encorafenib + Binimetinib, Surgery, Adjuvant Encorafenib + Binimetinib
Started | 3
Eligible and treated | 3
Completed | 1
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — No surgery within required timeframe due to Covid diagnosis | 1

BASELINE CHARACTERISTICS:
Population: All 3 patients enrolled are included in this analysis.
Arm/Group | Neoadjuvant Encorafenib + Binimetinib, Surgery, Adjuvant Encorafenib + Binimetinib
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 42 [31 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response
Description: Pathologic complete response (pCR) is defined as complete absence of viable tumor in the treated tumor bed. Partial pathologic response (pPR) is defined as less than or equal to 50% of the treated tumor bed is occupied by viable tumor cells. Pathologic non-response is defined as great than 50% of the treated tumor bed is occupied by viable tumor cells.
Time Frame: Assessed at 10-12 weeks
Population: All 3 enrolled patients are included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Encorafenib + Binimetinib, Surgery, Adjuvant Encorafenib + Binimetinib
Number analyzed (Participants) | 3
Participants
  Pathologic complete response | 2
  Pathologic partial response | 1

2. Secondary Outcome: Objective Response
Description: Objective response is defined as either complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Complete response is defined as disappearance of all lesions. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters and/or persistence of one or more non-target lesion(s). Stable disease is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Assessed at baseline, 8 weeks, then every 12 weeks up to 1.4 years
Population: All 3 enrolled patients are included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Encorafenib + Binimetinib, Surgery, Adjuvant Encorafenib + Binimetinib
Number analyzed (Participants) | 3
Participants
  partial response | 2
  stable disease | 1

3. Secondary Outcome: Disease-free Survival
Description: Disease-free survival is defined as the time from date of surgical resection to the date of recurrence or death, whichever occurs first.
  Recurrence must be documented by radiologic exams and with biopsy in all cases except for brain metastases (biopsy not required). Abnormal blood studies alone (e.g., elevated transaminases or alkaline phosphatase) are not sufficient evidence of relapse. Whenever possible, histologic proof of recurrence should be obtained unless the lesion is not accessible or a biopsy would cause undue risk to the patient.
Time Frame: Assessed at baseline, 8 weeks, then every 12 weeks up to 19.4 months
Population: All 3 patients enrolled were included.
Measure: Median (Full Range); unit: months
Arm/Group | Neoadjuvant Encorafenib + Binimetinib, Surgery, Adjuvant Encorafenib + Binimetinib
Number analyzed (Participants) | 3
months | 13.1 [8.3 to 19.4]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from registration to death or date last known alive, which is the censoring date for patients who are still alive.
Time Frame: Assessed at every 3 months for 2 years and then every 6 months, up to 2 years 9 months
Population: All 3 enrolled patients are included in this analysis. All 3 patients were alive as of this analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Neoadjuvant Encorafenib + Binimetinib, Surgery, Adjuvant Encorafenib + Binimetinib
Number analyzed (Participants) | 3
months | 24 [21.8 to 28.5]

5. Secondary Outcome: Associations Between pCR and Best Response
Description: Association between pCR and best response will be reported.
Time Frame: Assessed at baseline, 8 weeks, then every 12 weeks up to 1.4 years
Population: All enrolled patients are included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With pCR: Patients with pathologic complete response
- Patients Without pCR: Patients without pathologic complete response
Arm/Group | Patients With pCR | Patients Without pCR
Number analyzed (Participants) | 2 | 1
Participants
  Partial Response | 1 | 1
  Stable Disease | 1 | 0

6. Other Pre Specified Outcome: CD8+ T Cell Infiltration and Ki-67 Status
Description: Evaluation of CD8+ T cell infiltration and Ki-67 status in tumor or tumor bed pre, during, and post neoadjuvant treatment will be performed. The change in CD8+ TIL with neoadjuvant treatment will also be evaluated.
Time Frame: Assessed at baseline, during neoadjuvant treatment and at surgery
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Concordance Between Local Review for Pathologic Response and Central Pathology Review
Description: The concordance between local review for pathologic response and central pathology review will be performed.
Time Frame: Assessed at surgery
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in 18F-FLT PET/CT Uptake
Description: Comparison of the change in 18F-FLT PET/CT uptake from baseline to post-neoadjuvant therapy between patients with and without pathologic complete response will be performed.
Time Frame: Assessed at baseline and post-neoadjuvant therapy
Reporting Status: Not Posted

9. Other Pre Specified Outcome: 18F-FLT PET/CT Uptake
Description: The uptake value of 18F-FLT PET/CT will be evaluated after neoadjuvant treatment is completed. This value will be compared between patients with and without pathologic complete response.
Time Frame: Assessed after neoadjuvant treatment, about 16 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Association Between Pathologic Complete Response and Change in 18F-FLT PET/CT Uptake as Well as Post-neoadjuvant 18F-FLT PET/CT Uptake
Description: The association between pathologic complete response and change in 18F-FLT PET/CT uptake as well as post-neoadjuvant 18F-FLT PET/CT uptake will be evaluated. An optimal threshold of 18F-FLT PET/CT uptake for prediction of pathologic complete response will be estimated.
Time Frame: Assessed at baseline and post-neoadjuvant treatment
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Correlation Between Change in 18F-FLT PET/CT Uptake and Change in Ki-67
Description: The correlation between change in 18F-FLT PET/CT uptake and change in Ki-67 will be evaluated.
Time Frame: Assessed at baseline and post-neoadjuvant treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, up to 2 years and 9 months
Description: All 3 patients enrolled are included in the analysis of adverse events and all-cause mortality. As of this analysis, no patients had died.
Arm/Group | Experimental: Neoadjuvant Encorafenib + Binimetinib, Surgery, Adjuvant Encorafenib + Binimetinib
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Neoadjuvant Encorafenib + Binimetinib, Surgery, Adjuvant Encorafenib + Binimetinib (N=3)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Neoadjuvant Encorafenib + Binimetinib, Surgery, Adjuvant Encorafenib + Binimetinib (N=3)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Edema limbs (General disorders and administration site conditions) | 1
Fatigue (General disorders and administration site conditions) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Soft tissue infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
CPK increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT04221438/Prot_SAP_000.pdf